CLINICAL TRIAL: NCT06970821
Title: A Prospective Case-Control Study Investigating Serum Vitamin D Status and Metabolic Markers in Adolescent Girls With PCOS
Brief Title: Association of Vitamin D Status With Metabolic Markers in Adolescents With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nursen Kurtoglu Aksoy, Specialist in Obstetrics and Gynecology, Bagcilar Training and Research Hospital
Other Study IDs: 776/28.09.2023
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Polycystic Ovary Syndrome; Vitamin D Deficiency; Insulin Resistance
Keywords: Adolescents; Polycystic Ovary Syndrome; Metabolic Markers; Visceral fat
MeSH Terms: conditions — Polycystic Ovary Syndrome; Vitamin D Deficiency; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PCOS Group: Adolescents diagnosed with PCOS according to NIH criteria, evaluated for metabolic parameters and vitamin D status.
- Control Group: Healthy adolescents without PCOS, evaluated with the same clinical, biochemical, and ultrasound measures.

SUMMARY:
This prospective cross-sectional case-control study aims to investigate the relationship between serum vitamin D levels, visceral adipose tissue (VAT) thickness, and metabolic parameters in adolescents diagnosed with polycystic ovary syndrome (PCOS), compared to healthy controls. The study includes 70 adolescents with PCOS and 40 age-matched healthy adolescents, all aged between 12 and 19 years, who attended the adolescent gynecology outpatient clinic of a tertiary care hospital. Serum 25-hydroxy vitamin D [25(OH)D] levels, fasting glucose, fasting insulin, lipid profiles, anthropometric measurements, and ultrasound-based VAT thickness were assessed. The study seeks to explore potential associations between vitamin D deficiency and metabolic dysregulation in adolescent PCOS patients and to better understand the early cardiometabolic risks associated with PCOS during adolescence.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder affecting women of reproductive age, with manifestations often beginning during adolescence. It is associated not only with reproductive abnormalities but also with significant metabolic complications, including insulin resistance, obesity, dyslipidemia, and an increased risk of metabolic syndrome. Recent evidence suggests that vitamin D deficiency may play a role in the metabolic dysfunction observed in PCOS, although the exact mechanisms remain under investigation.

This prospective cross-sectional case-control study aims to evaluate the relationship between serum 25-hydroxy vitamin D [25(OH)D] levels, visceral adipose tissue (VAT) thickness, and metabolic parameters in adolescents with PCOS compared to healthy controls. The study population includes 70 adolescents diagnosed with PCOS according to the NIH criteria and 40 age-matched healthy adolescents, all aged between 12 and 19 years, attending a tertiary care hospital's adolescent gynecology clinic.

Participants underwent detailed clinical and anthropometric assessments, including measurements of body mass index (BMI), waist circumference, hip circumference, and waist-to-hip ratio (WHR). Biochemical evaluations included fasting plasma glucose, fasting insulin, lipid profiles, and serum 25(OH)D levels. Insulin resistance was assessed using the HOMA-IR .

VAT and subcutaneous adipose tissue (SAT) thickness were measured by transabdominal ultrasound, utilizing a standardized technique for consistency. All ultrasound measurements were performed by the same experienced investigator to ensure reliability, and intraobserver agreement was assessed.

The primary objective of the study is to investigate potential associations between vitamin D deficiency and metabolic disturbances in adolescents with PCOS, focusing particularly on insulin resistance, lipid abnormalities, and visceral fat accumulation. The findings may contribute to a better understanding of early cardiometabolic risk in adolescents with PCOS and help in developing targeted preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents aged 13 to 19 years
* Having attained menarche at least two years prior to enrollment
* For PCOS group: Diagnosis of polycystic ovary syndrome based on NIH criteria (presence of menstrual irregularity and clinical and/or biochemical hyperandrogenism)
* For Control group: Regular menstrual cycles (cycle interval 21-35 days) and no clinical or biochemical signs of hyperandrogenism.

Exclusion Criteria:

* Use of medications affecting vitamin D metabolism, insulin sensitivity, or androgen levels within the past 6 months (e.g., oral contraceptives, insulin sensitizers, vitamin D supplements)
* Presence of endocrine disorders such as congenital adrenal hyperplasia, hyperprolactinemia, Cushing's syndrome, thyroid dysfunction.
* Chronic systemic diseases (e.g., diabetes mellitus, severe liver or kidney disease).

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Female adolescents aged 13 to 19 years who attended the adolescent gynecology outpatient clinic of a tertiary care hospital. Participants included adolescents diagnosed with polycystic ovary syndrome based on NIH criteria and age-matched healthy controls. All participants had attained menarche at least two years prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Serum 25(OH)D Level at Baseline | At enrollment
  Concentration of 25-hydroxyvitamin D [25(OH)D] in serum measured in ng/mL using chemiluminescent immunoassay.
Body Mass Index (BMI) at Baseline | At enrollment
  Body mass index calculated as weight in kilograms divided by the square of height in meters (kg/m²).
HOMA-IR Value at Baseline | At enrollment
  Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) calculated as [fasting glucose (mg/dL) × fasting insulin (µU/mL)] / 405.
Serum Lipid Profile at Baseline | At enrollment
  Fasting serum levels of total cholesterol, HDL, LDL, and triglycerides measured in mg/dL.
Visceral Adipose Tissue Thickness, Subcutaneous Adipose Tissue Thickness | At enrollment
  The transducer was placed transversely, 1 cm above the umbilicus on the xiphoid-pubic line

CONTACTS AND LOCATIONS:
Overall Officials: Nese Hayirlioglu, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bağcılar Training and Research Hospital, Istanbul, Turkey (Türkiye)